CLINICAL TRIAL: NCT00901017
Title: A Randomised Controlled Spilt-mouth Clinical Study Comparing a Synthetic Bone Substitute and a Bovine-derived Xenograft in Primarily Horizontal Bone Augmentation Procedure During Placement of Straumann Oral Implants
Brief Title: Comparison of Synthetic Bone Substitute and a Bovine-derived Xenograft in Horizontal Bone Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 04/05
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Jaw, Edentulous; Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous; Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Straumann BoneCeramic (Active Comparator): Straumann BoneCeramic
  Interventions: Device: Straumann BoneCeramic
- Bio-Oss (Active Comparator): Geistlich Bio-Oss
  Interventions: Device: Bio-Oss

INTERVENTIONS:
Device: Straumann BoneCeramic — Bone augmentation procedure performed with Bone Ceramic
  Arms: Straumann BoneCeramic
Device: Bio-Oss — Bone Augmentation procedure performed with Bio Oss
  Arms: Bio-Oss

SUMMARY:
The objective of the study is to test the efficacy on bone formation of Straumann Bone Ceramic as a grafting material applied in buccal bone dehiscences on simultaneously placed oral implants.

DETAILED DESCRIPTION:
This is a randomized, controlled, split mouth, prospective, single centre study. The total study duration for each patient should be 76 weeks +/-18 months.

In total 8 visits per patient are scheduled in this study.

The study devices Straumann Bone Ceramic and Bio-Oss are CE-marked, and approved by the FDA. The products are used within the indication.

One center in Beligum will participate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years to 80 years of age
* At least two missing teeth up to full edentulous arches.
* Desiring implant supported restorations.
* Both study implants should have a self-containing (2-wall) buccal dehiscence defect after oral implant placement (at least 3.0 mm / max. 5.0 mm defect in apico-coronal aspect to be measured from the boarder of the rough surface of the oral implant to the bottom of the defect).
* At least 4mm of the implant, measured from the apical end to the lowest margin of the bone level, should be covered with bone.
* Sufficient bone volume such that both oral implants will not encroach on vital structures and primary stability of the oral implant can be achieved;
* Patients must be committed to the study and must sign informed consent.
* Patient in good general health as documented by self assessment;
* Full mouth plaque score of <20%;

Exclusion Criteria:

* Any systemic medical condition that could interfere with the surgical procedure or planned treatment;
* Current pregnancy or breast feeding/ lactating at the time of recruitment;
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene;
* Alcoholism or chronically drug abuse causing systemic compromise.
* Patients who smoke more than 20 cigarettes per day.
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for surgical procedure or would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability
* Lack of primary stability of 1 or both implant(s) at surgery, measured by hand testing. In this instance the patient must be withdrawn and treated accordingly.
* Mucosal diseases such as erosive lichen planus
* History of local radiation therapy.
* Presence of osseous pathologies.
* Presence of oral lesions (such as ulceration, malignancy)
* Severe bruxing or clenching habits.
* Local inflammation, including untreated periodontitis.
* Bone surgery at the implant site(s) (bone grafts, guided tissue regeneration techniques for bone enhancement) prior to implant placement unless performed more than 6 months prior to implant placement.
* Patients presenting clinical and radiological signs and symptoms of maxillary sinus disease.
* Existing teeth in the residual dentition with untreated endodontic pathologies.
* Patients with inadequate oral hygiene or unmotivated for adequate home care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quirynen, Professor, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Straumann BoneCeramic and Geistlich Bio-Oss: Each patient received both treatments in a split-mouth design.
Period: Overall Study
Arm/Group | Straumann BoneCeramic and Geistlich Bio-Oss
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Straumann BoneCeramic and Geistlich Bio-Oss
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 14

OUTCOME MEASURES:

1. Primary Outcome: Change of Vertical Height of Buccal Defects
Description: Change of vertical height of buccal defects over 26 weeks, measured during 1st - and 2nd- stage surgery
Time Frame: Baseline to 26 weeks
Population: 14 patients represented the ITT population.
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Straumann BoneCeramic: In the test site the bone grafting procedure will be done with a synthetic biphasic calcium phosphate in particulate form (Straumann Bone Ceramic, Institute Straumann AG, Switzerland).
- Geistlich Bio-Oss: The control site will be treated with a granular bone substitute derived from bovine bone (Bio-Oss - Geistlich Biomaterials, Wollhusen, Switzerland).
Arm/Group | Straumann BoneCeramic | Geistlich Bio-Oss
Number analyzed (Participants) | 14 | 14
mm | -4.5 [-5.8 to -3.2] | -4.82 [-5.9 to -3.7]

2. Secondary Outcome: Implant Success Rate
Description: The success of oral implant will be determined according to the following parameters:
  * Absence of any continuous peri-implant radiolucency based on radiographic findings.
  * Absence of implant mobility (based on hand testing)
  * Absence of a peri-implant infection with suppuration.
  * Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if it is observed at two or more follow-up visits after treatment with systemic antibiotics).
  * Bone level changes evaluated on periapical radiographs around implants less than 1 mm during the first year of loading, starting at abutment connection.
Time Frame: 6 months
Measure: Number; unit: % of implants
Arm/Group | Straumann BoneCeramic | Geistlich Bio-Oss
Number analyzed (Participants) | 14 | 14
% of implants | 100 | 100

3. Secondary Outcome: Implant Survival Rate
Description: A surviving implant will be considered an implant fulfilling the following criteria:
  * Absence of any continuous peri-implant radiolucency based on radiographic findings.
  * Absence of implant mobility.
  * Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if it is observed at two or more follow-up visits after treatment with systemic antibiotics).
  * Absence of pain or any other adverse observation by the patient, so that the implant has to be removed.
Time Frame: 6 Months
Measure: Number; unit: % of implants
Arm/Group | Straumann BoneCeramic | Geistlich Bio-Oss
Number analyzed (Participants) | 14 | 14
% of implants | 100 | 100

4. Secondary Outcome: Implant Success Rate
Description: as for outcome 2
Time Frame: 12 months
Measure: Number; unit: % of implants
Arm/Group | Straumann BoneCeramic | Geistlich Bio-Oss
Number analyzed (Participants) | 14 | 14
% of implants | 100 | 100

5. Secondary Outcome: Implant Survival Rate
Description: as for outcome 3
Time Frame: 12 months
Measure: Number; unit: % of implants
Arm/Group | Straumann BoneCeramic | Geistlich Bio-Oss
Number analyzed (Participants) | 14 | 14
% of implants | 100 | 100

ADVERSE EVENTS:
Arm/Group | Straumann BoneCeramic | Geistlich Bio-Oss
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Straumann BoneCeramic (N=14) | Geistlich Bio-Oss (N=14)
Membrane necrosis (General disorders) | 1 (1) | 1 (1)
Perforation (General disorders) | 1 (1) | 1 (1)
Candida (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days